CLINICAL TRIAL: NCT03198078
Title: A Multicenter, Randomized, Double-blind, Placebo- and Active-controlled Trial to Evaluate the Efficacy of Brexpiprazole Monotherapy for the Treatment in Adolescents (13-17 Years Old) With Schizophrenia
Brief Title: Trial to Evaluate the Short-term Safety & Efficacy of Brexpiprazole Monotherapy in the Treatment of Adolescents With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-10-234; 2017-001447-12 (EudraCT Number)
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia
Keywords: Brexpiprazole; Schizophrenia; Adolescent
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole; Aripiprazole

STUDY DESIGN:
Intervention Model Description: Subjects randomized 1:1:1 to 1 of 3 double-blind treatment arms to evaluate safety & efficacy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brexpiprazole (Experimental): Participants were administered with brexpiprazole oral tablets, daily, dose titrated up to 0.5 mg by Day 4, 1 mg by Day 7, 2 mg by Day 14, then between 2-4 mg after Day 21 up to Week 6 with a 1 mg increase or decrease, based on the Investigator's decision.
  Interventions: Drug: Brexpiprazole (OPC-34712)
- Aripiprazole (Active Comparator): Participants were administered with aripiprazole oral tablets, daily, dose titrated up to 2 mg by Day 4, 5 mg by Day 7, 10 mg by Day 14, then 10, 15 or 20 mg after Day 21 up to Week 6 with a 5 mg increase or decrease, based on the Investigator's decision.
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): Participants were administered with brexpiprazole or aripiprazole matching placebo oral tablets, daily up to Week 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole (OPC-34712) — Once-daily, tablets
  Arms: Brexpiprazole
Drug: Aripiprazole — Once-daily, tablets
  Arms: Aripiprazole
Drug: Placebo — Once-daily, tablets
  Arms: Placebo

SUMMARY:
To determine the safety & efficacy of brexpiprazole monotherapy in the treatment of adolescents with schizophrenia.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo- and active-controlled trial to evaluate the safety and efficacy of brexpiprazole monotherapy compared to placebo in adolescent subjects (ages 13-17) with a DSM-5 diagnosis of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male & female subjects aged 13-17 years, inclusive at time of consent and at baseline visit, with a primary diagnosis of schizophrenia as defined by DSM-5 criteria and confirmed by K-SADS-PL and a history of the illness for at least 6 months prior to screening.
* PANSS score >= 80, inclusive, at screening and baseline

Exclusion Criteria:

* Subjects with a DSM-5 diagnosis other than schizophrenia that has been the primary focus of treatment within 3 months of screening.
* Subjects with a clinical presentation or history that is consistent with delirium, dementia, amnesia or other cognitive disorders
* Subjects who have been hospitalized > 21 days for a current exacerbation of schizophrenia at the time of baseline.
* Any neurological disorder other than Tourette's Syndrome
* Subjects at significant risk of committing violent acts, serious self-harm or suicide based on history
* Subjects with epilepsy, a history of seizures, severe head trauma or stroke
* Subjects who test positive for drugs of abuse at screening

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Ward, PhD., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Ward C, Pejovic Milovancevic M, Kohegyi E, Hefting N, Aurang C, Chen D, Larsen KG, Hobart M, Correll CU. Efficacy and safety of brexpiprazole in adolescents with schizophrenia: a multicountry, randomised, double-blind, placebo-controlled, phase 3 trial with an active reference. Lancet Psychiatry. 2025 May;12(5):345-354. doi: 10.1016/S2215-0366(25)00043-4. Epub 2025 Apr 7. PMID 40209740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigational sites in the United States, Mexico, France, Italy, Poland, Romania, Serbia, Spain, Ukraine, and Russia from 30 June 2017 to 03 April 2023.
Pre-assignment Details: A total of 376 participants were screened, of which 316 participants were enrolled and randomized to brexpiprazole, aripiprazole or placebo groups in 1:1:1 ratio.
Period: Overall Study
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Started | 110 | 102 | 104
Safety Sample (Safety sample included all randomized participants who received at least 1 dose of investigational medicinal product (IMP).) | 110 | 102 | 104
Efficacy Sample (Efficacy sample included all randomized participants who received at least 1 dose of IMP, had a baseline assessment, and at least one post-baseline assessment of the Positive and Negative Syndrome Scale (PANSS) Total Score.) | 110 | 101 | 103
Completed | 107 | 97 | 92
Not Completed | 3 | 5 | 12
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Withdrawal by Caregiver | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Randomized sample included all participants who were randomized into the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 110 | 102 | 104 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.5) | 15.3 (1.4) | 15.2 (1.4) | 15.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 57 | 51 | 166
  Male | 52 | 45 | 53 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 70 | 66 | 68 | 204
  Race: Black or African American | 8 | 7 | 6 | 21
  Race: American Indian or Alaska Native | 2 | 1 | 4 | 7
  Race: Asian | 1 | 1 | 0 | 2
  Race: Other | 29 | 27 | 25 | 81
  Race: Missing | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 34 | 32 | 34 | 100
  Ethnicity: Not Hispanic or Latino | 75 | 70 | 68 | 213
  Ethnicity: Other | 1 | 0 | 1 | 2
  Ethnicity: Missing | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 14 | 43
  France | 0 | 0 | 1 | 1
  Italy | 1 | 1 | 1 | 3
  Mexico | 32 | 31 | 32 | 95
  Poland | 5 | 3 | 3 | 11
  Romania | 6 | 6 | 6 | 18
  Russia | 4 | 4 | 3 | 11
  Serbia | 11 | 10 | 10 | 31
  Spain | 1 | 0 | 0 | 1
  Ukraine | 35 | 33 | 34 | 102
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) to 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranges from 30 (best possible outcome) to 210 (worst possible outcome). Higher scores indicate worsening of symptoms.
  score on a scale | 101.1 (14.9) | 101.0 (13.0) | 102.1 (16.3) | 101.4 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) to 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranges from 30 (best possible outcome) to 210 (worst possible outcome). Higher scores indicate worsening of symptoms. Least squares (LS) mean was determined by Mixed-effect model repeated measures (MMRM) method with fixed effect of treatment, (pooled) clinical center visit, treatment visit interaction, baseline value and baseline visit interaction as a covariate, and with an unstructured covariance.
Time Frame: Baseline to Week 6
Population: Efficacy sample included all randomized participants who received at least 1 dose of IMP, had a baseline assessment, and at least one post-baseline assessment of the PANSS Total Score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale | -22.75 (1.49) | -23.95 (1.57) | -17.42 (1.58)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.0136, MMRM — P-value was analyzed by MMRM method with fixed effect of treatment, (pooled) clinical center visit, treatment visit interaction, baseline value, and baseline visit interaction as a covariate, and with an unstructured covariance; LS mean difference = -5.33, 95% CI 2-sided [-9.55 to -1.10]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; p = 0.0032, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -6.53, 95% CI 2-sided [-10.8 to -2.21]

2. Secondary Outcome: Change From Baseline to Week 6 in PANSS Positive and Negative Sub-Scales Scores
Description: PANSS has 7 positive symptom constructs: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility; and 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. Each item's severity was rated on 7-point scale, with score of 1 (absence of symptoms) to 7 (extremely severe symptoms). PANSS positive & negative subscale scores were the sum of rating scores for 7 positive & 7 negative items respectively. Both scores range from 7 (best possible outcome) to 49 (worst possible outcome). Higher scores denote worsening of symptoms. LS mean was determined by MMRM method with fixed effect of treatment, (pooled) clinical center visit, treatment visit interaction, baseline value, and baseline visit interaction as a covariate, and with an unstructured covariance.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale
  Change From Baseline to Week 6 in PANSS Positive Sub-scale Score | -6.58 (0.43) | -7.29 (0.45) | -5.14 (0.46)
  Change From Baseline to Week 6 in PANSS Negative Sub-scale Score | -4.70 (0.41) | -4.77 (0.43) | -3.82 (0.44)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Change From Baseline to Week 6 in PANSS Positive Sub-scale Score; Test type: Superiority; p = 0.0205, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -1.44, 95% CI 2-sided [-2.65 to -0.22]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Change From Baseline to Week 6 in PANSS Positive Sub-scale Score; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -2.15, 95% CI 2-sided [-3.40 to -0.91]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Change From Baseline to Week 6 in PANSS Negative Sub-scale Score; Test type: Superiority; p = 0.1360, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.88, 95% CI 2-sided [-2.04 to 0.28]
Statistical Analysis 4: Comparison: Aripiprazole vs Placebo; Change From Baseline to Week 6 in PANSS Negative Sub-scale Score; Test type: Superiority; p = 0.1158, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.95, 95% CI 2-sided [-2.14 to 0.24]

3. Secondary Outcome: Percentage of Participants Achieving Response
Description: Response was defined as at least 30% improvement from baseline in PANSS Total Score or CGI score of 1 or 2. The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel, and ranges from 30 (best possible outcome) to 210 (worst possible outcome). The CGI scale is an investigator-rated evaluation that assesses the severity of a participant's illness on a 7-point scale, ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Percentage of participants achieving response was determined by Last Observation Carried Forward (LOCF) method.
Time Frame: Up to 6 weeks
Population: Efficacy sample included all randomized participants who received at least 1 dose of IMP, had a baseline assessment, and at least one post-baseline assessment of the PANSS Total Score. Percentages are rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
percentage of participants | 43.64 | 43.56 | 28.16
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.0111, Cochran-Mantel-Haenszel; P-value was analyzed by Cochran-Mantel-Haenszel (CMH) general association test controlling for (pooled) centers; Ratio of Response Rate = 1.55, 95% CI 2-sided [1.09 to 2.20]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; p = 0.0224, Cochran-Mantel-Haenszel; P-value was analyzed by CMH general association test controlling for (pooled) centers; Ratio of Response Rate = 1.51, 95% CI 2-sided [1.06 to 2.16]

4. Secondary Outcome: Percentage of Participants Achieving Remission
Description: Remission was defined as a score of ≤ 3 on each of the following specific PANSS items: delusions (positive scale item [P] 1), unusual thought content (general scale item [G] 9), hallucinatory behavior (P3), conceptual disorganization (P2), mannerisms/posturing (G5), blunted affect (negative scale item [N] 1), passive/apathetic social withdrawal (N4), and lack of spontaneity and conversation flow (N6). Each item's severity was rated on 7-point scale, with score of 1 (absence of symptoms) to 7 (extremely severe symptoms). Percentage of participants achieving remission was determined by LOCF method.
Time Frame: Up to 6 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
percentage of participants | 29.09 | 35.64 | 23.30
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.4415, Cochran-Mantel-Haenszel; P-value was analyzed by CMH general association test controlling for (pooled) centers; Ratio of Remission Rate = 1.18, 95% CI 2-sided [0.77 to 1.81]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; p = 0.0472, Cochran-Mantel-Haenszel; P-value was analyzed by CMH general association test controlling for (pooled) centers; Ratio of Remission Rate = 1.48, 95% CI 2-sided [1.01 to 2.16]

5. Secondary Outcome: Change From Baseline to Week 6 in Children's Global Assessment Scale (CGAS) Total Score
Description: The CGAS is a 100-point rating scale measuring psychological, social, and school functioning for children aged 6-17 years and provides a global measure of the severity of disturbance. The scale is separated into 10-point sections that are headed with a description of the level of functioning and followed by examples matching the interval. The score ranges from 0-100, 1 to 10 indicates the need for constant supervision and 91 to 100 indicates superior functioning in all areas. Higher scores indicate better functioning. LS mean was determined by MMRM method with fixed effect of treatment, (pooled) clinical center visit, treatment visit interaction, baseline value, and baseline visit interaction as a covariate, and with an unstructured covariance.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale | 10.56 (1.00) | 12.07 (1.05) | 8.08 (1.06)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.0854, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 2.48, 95% CI 2-sided [-0.35 to 5.31]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; p = 0.0072, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 3.99, 95% CI 2-sided [1.09 to 6.88]

6. Secondary Outcome: Change From Baseline to Week 6 in Clinical Global Impression Severity (CGI-S) Scale Score
Description: The CGI-S scale is an investigator-rated evaluation that assesses the severity of a participant's illness on a 7-point scale, ranging from 1 to 7. The investigator answered the question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?". Response choices were: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. Higher scores indicate worse condition. LS mean was determined by the MMRM method with fixed effect of treatment, (pooled) clinical center visit, treatment visit interaction, baseline value, and baseline visit interaction as a covariate, and with an unstructured covariance.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale | -0.92 (0.09) | -1.01 (0.09) | -0.80 (0.09)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.3589, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.11, 95% CI 2-sided [-0.36 to 0.13]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; p = 0.1118, MMRM — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.20, 95% CI 2-sided [-0.45 to 0.05]

7. Secondary Outcome: Mean Clinical Global Impression Improvement (CGI-I) Scale Score at Week 6
Description: The efficacy of brexpiprazole in the treatment was rated for each participant using the CGI-I. The investigator rated the participant's total improvement whether or not it was entirely due to drug treatment on a 7-point scale, ranging from 0 to 7. Response choices were: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Higher scores indicate worse condition. Mean CGI-I scale score was determined by LOCF method.
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale | 2.86 (0.95) | 2.79 (0.97) | 3.17 (1.08)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.0287, Cochran-Mantel-Haenszel; P-value was analyzed by CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.56 to -0.03]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; p = 0.0184, Cochran-Mantel-Haenszel; P-value was analyzed by CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.62 to -0.06]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Trial Discontinuation Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered with a medicinal product that does not necessarily have a causal relationship with the treatment.
Time Frame: From the first dose of study drug up to 21 days after the last dose of study drug (up to approximately 9 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 102 | 104
Participants
  AEs | 46 | 56 | 44
  Trial Discontinuation Due to AEs | 0 | 1 | 2

9. Secondary Outcome: Number of Participants With Treatment-emergent AEs (TEAEs), Serious TEAEs, and TEAEs Graded by Severity
Description: An AE was defined as any untoward medical occurrence in a participant administered with a medicinal product that does not necessarily have a causal relationship with the treatment. An SAE was any AE that results in the appearance of (or worsening of any pre-existing) undesirable signs, symptoms, or medical conditions which is fatal, life-threatening, result in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, and requires inpatient hospitalization or prolongation of existing hospitalization. TEAE is any AE after the start of treatment or if the event was continuous from baseline, medicinal product related, or resulted in death, discontinuation, interruption or reduction of medicinal product. TEAEs were graded on a 3-point scale: 1 (Mild: Discomfort noticed, but no disruption to daily activity), 2 (Moderate: Discomfort sufficient to reduce or affect normal daily activity), and 3 (Severe: Inability to work or perform normal daily activity).
Time Frame: From the first dose of study drug up to 21 days after the last dose of study drug (up to approximately 9 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Brexpiprazole 2 to 4 mg/Day: Participants were administered with brexpiprazole oral tablets, daily, dose titrated up to 0.5 mg by Day 4, 1 mg by Day 7, 2 mg by Day 14, then between 2-4 mg after Day 21 up to Week 6 with a 1 mg increase or decrease, based on the Investigator's decision.
- Aripiprazole 10 to 20 mg/Day: Participants were administered with aripiprazole oral tablets, daily, dose titrated up to 2 mg by Day 4, 5 mg by Day 7, 10 mg by Day 14, then 10, 15 or 20 mg after Day 21 up to Week 6 with a 5 mg increase or decrease, based on the Investigator's decision.
Arm/Group | Brexpiprazole 2 to 4 mg/Day | Aripiprazole 10 to 20 mg/Day | Placebo
Number analyzed (Participants) | 110 | 102 | 104
Participants
  TEAEs | 44 | 53 | 42
  Serious TEAEs | 1 | 1 | 3
  Mild TEAEs | 33 | 47 | 32
  Moderate TEAEs | 17 | 16 | 13
  Severe TEAEs | 2 | 0 | 1

10. Secondary Outcome: Mean Change From Baseline in Weight
Description: Change in weight was reported, in kilograms (kg).
Time Frame: Baseline up to last visit (approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
kg | 0.8 (2.6) | 0.5 (2.7) | 0.0 (2.2)

11. Secondary Outcome: Mean Change From Baseline in Height
Description: Change in height was reported in centimeters (cm).
Time Frame: Baseline up to last visit (approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with data available for the outcome measure analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 108 | 99 | 96
cm | 0.2 (1.1) | 0.2 (2.9) | 0.3 (0.6)

12. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI)
Description: Change in BMI was reported in kilograms per square meter (kg/m^2).
Time Frame: Baseline up to last visit (approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed indicates the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 108 | 99 | 96
kg/m^2 | 0.2 (1.1) | 0.3 (1.5) | 0.0 (0.9)

13. Secondary Outcome: Mean Change From Baseline in Waist Circumference
Description: Change in waist circumference was reported in 'cm'.
Time Frame: Baseline up to last visit (approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
cm | 0.6 (3.9) | -0.3 (4.3) | 0.0 (5.1)

14. Secondary Outcome: Number of Participants With At Least One Occurrence of Suicidal Behavior or Suicidal Ideation as Recorded on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a scale used to report at least one occurrence of any suicidal behavior or suicidal ideation. Suicidal behavior was defined as reporting any of the following items: actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior. The suicidal ideation total score is the sum of intensity scores of 5 items (frequency, duration, controllability, deterrents, and reasons for ideation). The score of each intensity item ranges from 0 (none) to 5 (worst) and the total score ranges from 0 to 25. Lower scores indicate improvement.
Time Frame: From the first dose of study drug up to last dose of study drug (up to approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 102 | 104
Participants | 1 | 2 | 2

15. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Test Values
Description: Potentially clinically relevant laboratory values assessed included - serum chemistry [including blinded prolactin], hematology, and urinalysis as defined in SAP.
Time Frame: From the first dose of study drug up to last dose of study drug (up to approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with data available for the outcome measure analysis. 'Number analyzed' indicates the number of participants with at least one post-baseline numeric result for the specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 105 | 98 | 99
Participants
  Alanine Aminotransferase (U/L): High: number analyzed (Participants) | 105 | 98 | 98
  Alanine Aminotransferase (U/L): High | 1 | 2 | 0
  Bilirubin (mg/dL): High: number analyzed (Participants) | 105 | 96 | 91
  Bilirubin (mg/dL): High | 0 | 1 | 0
  Cholesterol, Fasting (mg/dL): High: number analyzed (Participants) | 102 | 98 | 96
  Cholesterol, Fasting (mg/dL): High | 2 | 3 | 0
  Creatine kinase (U/L): High: number analyzed (Participants) | 105 | 98 | 98
  Creatine kinase (U/L): High | 5 | 4 | 1
  Glucose, Fasting (mg/dL): High: number analyzed (Participants) | 102 | 98 | 96
  Glucose, Fasting (mg/dL): High | 16 | 15 | 9
  HDL Cholesterol, Fasting (mg/dL): Low: number analyzed (Participants) | 100 | 96 | 94
  HDL Cholesterol, Fasting (mg/dL): Low | 12 | 10 | 13
  LDL Cholesterol, Fasting (mg/dL): High: number analyzed (Participants) | 100 | 96 | 94
  LDL Cholesterol, Fasting (mg/dL): High | 2 | 3 | 0
  Triglycerides, Fasting (mg/dL): High: number analyzed (Participants) | 102 | 98 | 96
  Triglycerides, Fasting (mg/dL): High | 13 | 7 | 10
  Urate (mg/dL): High: number analyzed (Participants) | 105 | 98 | 98
  Urate (mg/dL): High | 0 | 0 | 1
  Eosinophils/Leukocytes (%): High: number analyzed (Participants) | 104 | 98 | 99
  Eosinophils/Leukocytes (%): High | 2 | 0 | 0
  Hematocrit (%): Low: number analyzed (Participants) | 104 | 97 | 98
  Hematocrit (%): Low | 4 | 0 | 1
  Hemoglobin (g/dL): Low: number analyzed (Participants) | 104 | 98 | 99
  Hemoglobin (g/dL): Low | 2 | 0 | 0
  Leukocytes (10^9/L): Low: number analyzed (Participants) | 104 | 98 | 99
  Leukocytes (10^9/L): Low | 0 | 1 | 0
  Leukocytes (10^9/L): High: number analyzed (Participants) | 104 | 98 | 99
  Leukocytes (10^9/L): High | 0 | 0 | 1
  Protein, Urine: High: number analyzed (Participants) | 105 | 98 | 97
  Protein, Urine: High | 2 | 2 | 0

16. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Abnormalities in Vital Signs
Description: Vital sign measurements included body weight, systolic blood pressure (SBP), and diastolic blood pressure (DBP). Blood pressure measurements were made in the supine, sitting, and standing positions after the participant had been in each position for at least 3 minutes as defined in SAP.
Time Frame: From the first dose of study drug up to last dose of study drug (up to approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with at least one post-baseline result for the specified vital signs.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
Participants
  SBP Sitting (mmHg): Low | 0 | 0 | 1
  SBP Standing (mmHg): Low | 1 | 1 | 0
  SBP Supine (mmHg): Low | 0 | 0 | 1
  DBP Standing (mmHg): Low | 1 | 0 | 0
  DBP Supine (mmHg): Low | 0 | 1 | 0
  Weight (kg): Low | 5 | 2 | 4
  Weight (kg): High | 9 | 5 | 5
  Orthostatic Hypotension (mmHg): Low | 2 | 1 | 2

17. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Parameters
Description: Twelve-lead ECG recordings were obtained after the participant was supine and at rest for at least 5 minutes as defined in SAP.
Time Frame: From the first dose of study drug up to last dose of study drug (up to approximately 6 weeks)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 107 | 97 | 94
Participants
  Rate: Bradycardia: number analyzed (Participants) | 107 | 97 | 93
  Rate: Bradycardia | 0 | 0 | 1
  Rhythm: Sinus Bradycardia: number analyzed (Participants) | 107 | 97 | 93
  Rhythm: Sinus Bradycardia | 0 | 0 | 1
  Rhythm: Supraventricular Premature Beat | 0 | 1 | 1
  Rhythm: Ventricular Premature Beat: number analyzed (Participants) | 106 | 97 | 93
  Rhythm: Ventricular Premature Beat | 1 | 0 | 0
  ST/T Morphology: QTcF: number analyzed (Participants) | 107 | 97 | 93
  ST/T Morphology: QTcF | 0 | 1 | 0
  ST/T Morphology: QTcN: number analyzed (Participants) | 107 | 97 | 93
  ST/T Morphology: QTcN | 0 | 1 | 0

18. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score
Description: The SAS consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Severity of each item was rated on a 5-point scale, with a score of 0 (absence of symptoms) to 4 (severe condition). The SAS total score is the sum of the scores of all 10 items, ranging from 0 to 40 where lower scores indicate less severe condition. LS mean was determined by Analysis of Covariance (ANCOVA) model with treatment and study center as main effects and baseline value as covariate.
Time Frame: Baseline up to last visit (approximately 6 weeks)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale | 0.04 (0.12) | 0.15 (0.12) | -0.03 (0.13)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; LS mean difference = 0.07, 95% CI 2-sided [-0.24 to 0.39] — LS mean difference was analyzed by ANCOVA model, with treatment and study center as main effects and baseline value as covariate
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; LS mean difference = 0.18, 95% CI 2-sided [-0.14 to 0.51] — [estimate comment as in outcome 18, analysis 1]

19. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS assessment consists of 12 items rating the involuntary movements: Facial and oral movements (4 items), extremity movements (2 items), and trunk movements (1 item) were observed unobtrusively while the participant is at rest and the investigator also made global judgments on the participant's dyskinesias (2 items), and dental status (2 items). Severity of each item was rated on a 5-point scale, with a score of 0 (absence of symptoms) to 4 (severe condition). Total Score is the sum of the scores of all 12 items, ranging from 0 to 48, higher scores indicate severe condition. LS mean was determined by ANCOVA model with treatment and study center as main effects and baseline value as covariate.
Time Frame: Baseline up to last visit (approximately 6 weeks)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale | -0.12 (0.09) | 0.05 (0.09) | -0.06 (0.09)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; LS mean difference = -0.06, 95% CI 2-sided [-0.30 to 0.18] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; LS mean difference = 0.11, 95% CI 2-sided [-0.13 to 0.36] — [estimate comment as in outcome 18, analysis 1]

20. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Score
Description: The BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the participant, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items were rated on a 4-point scale, with a score of 0 (absence of symptoms) to 3 (severe condition) and the global clinical assessment was rated on a 6-point scale, with a score of 0 (absence of symptoms) to 5 (severe akathisia). Total score is the sum of the scores of all 4 items, ranging from 0 to 14, higher scores indicate severe condition. LS mean was determined by ANCOVA model with treatment and study center as main effects and baseline value as covariate.
Time Frame: Baseline up to last visit (approximately 6 weeks)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 101 | 103
score on a scale | 0.01 (0.03) | 0.06 (0.03) | 0.01 (0.03)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; LS mean difference = 0.00, 95% CI 2-sided [-0.08 to 0.09] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Aripiprazole vs Placebo; Test type: Superiority; LS mean difference = 0.05, 95% CI 2-sided [-0.04 to 0.14] — [estimate comment as in outcome 18, analysis 1]

21. Secondary Outcome: Number of Participants With Severe Psychotropic Side Effects as Assessed by Udvalg for Kliniske Undersogelser (UKU) Rating Scale
Description: The UKU rating scale is a semi-structured interview used to assess the side effects of participants being treated with antipsychotic drugs. The scale is divided into 6 sub-scales: Psychic, neurological, autonomic, other, global assessment by subject, and global assessment by doctor. The scale has a total of 48 items, each item is rated on a 4-point scale (0=not present; 1=mild; 2=moderate; 3=severe), and the total score ranges from 0 to 144. Higher ratings indicate greater impairment. The severe side effects are reported in this outcome measure.
Time Frame: From the first dose of study drug up to last dose of study drug (up to approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 102 | 104
Participants
  Psychic: Concentration Difficulties | 7 | 10 | 8
  Psychic: Asthenia/Lassitude | 6 | 3 | 1
  Psychic: Failing Memory | 2 | 2 | 4
  Psychic: Depression | 0 | 2 | 1
  Psychic: Tension/Inner Unrest | 4 | 3 | 9
  Psychic: Increased Duration of Sleep | 0 | 1 | 0
  Psychic: Reduced Duration of Sleep | 4 | 1 | 1
  Psychic: Increased Dream Activity | 0 | 2 | 0
  Psychic: Emotional Indifference | 3 | 6 | 6
  Neurologic: Akathisia | 1 | 1 | 0
  Autonomic: Nausea/Vomiting | 0 | 0 | 1
  Autonomic: Micturition Disturbances | 0 | 1 | 0
  Autonomic: Palpitations/Tachycardia | 1 | 0 | 1
  Autonomic: Increased Tendency to Sweating | 1 | 0 | 0
  Other: Weight Gain | 0 | 1 | 0
  Other: Amenorrhoea | 0 | 1 | 0
  Other: Migraine | 0 | 0 | 1

22. Secondary Outcome: Number of Participants With Cognitive Adverse Effects Assessed by New York Assessment for Adverse Cognitive Effects of Neuropsychiatric Treatment (NY-AACENT)
Description: The NY-AACENT is used to detect changes in cognitive function subsequent to pharmacological or similar treatments for neurological or psychiatric problems, specifically designed to be used in pediatric population (ages 12 to 17), but could have been utilized with other age groups, as appropriate. Number of participants with at least one occurrence of the corresponding signs/symptoms are reported in this outcome measure.
Time Frame: From the first dose of study drug up to last dose of study drug (up to approximately 6 weeks)
Population: Safety sample included all randomized participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
Number analyzed (Participants) | 110 | 102 | 104
Participants
  Working Memory | 88 | 79 | 83
  Attention/Vigilance | 98 | 90 | 91
  Verbal Learning | 71 | 70 | 69
  Visual Learning | 46 | 46 | 44
  Reasoning | 97 | 86 | 83
  Speed of Processing | 88 | 84 | 82
  Social Cognition | 91 | 87 | 84
  Any Signs/Symptoms | 100 | 91 | 92

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 21 days after the last dose of study drug (up to approximately 9 weeks)
Description: Safety sample included all randomized participants who received at least 1 dose of IMP.
Arm/Group | Brexpiprazole | Aripiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/102 | 0/104
Serious Adverse Events (participants affected / at risk) | 1/110 | 1/102 | 3/104
Other Adverse Events (participants affected / at risk) | 19/110 | 28/102 | 16/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=110) | Aripiprazole (N=102) | Placebo (N=104)
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=110) | Aripiprazole (N=102) | Placebo (N=104)
Nausea (Gastrointestinal disorders) | 7 | 4 | 4
Fatigue (General disorders) | 2 | 8 | 0
Akathisia (Nervous system disorders) | 4 | 7 | 3
Headache (Nervous system disorders) | 7 | 5 | 5
Somnolence (Nervous system disorders) | 5 | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03198078/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT03198078/SAP_001.pdf